

## Centre for Clinical Vaccinology and Tropical Medicine University of Oxford, Churchill Hospital Headington, Oxford, OX3 7LE

**Title of Project:** Investigating the Impact of the Pulmonary Innate Immune Response and microbiome after exposure to Mycobacterium Tuberculosis – LIMBO-TB

**Researchers:** Helen McShane, Timothy Fredsgaard-Jones

| REC | ref: 24/EE/0070 IRAS ref: 337148 | | Please | Initial |
|---|---|---|---|---|
| 1. | I confirm that I have read and understand the Participant Information Sheet version, dated, for the above study. I have had the opportunity to consider the information, ask questions and these have been answered satisfactorily. | | | |
| 2. | I understand that I am free to withdraw at any time, without giving any reason, without my regal rights being affected. I understand that it may not be possible to destroy samples or respreviously gifted if they have already been used. | | | |
| 3. | I agree that relevant sections of my medical notes and data collected during the study can be responsible individuals from the University of Oxford, the National Health Service, study mor regulatory authorities, where it is relevant to my taking part in this research. I give permissio individuals to have access to my records. | nitors and | | |
| 4. | I agree that my GP can be informed of my participation, and I permit my GP to share my med with the research team if requested | lical history | | |
| 5. | I understand that the samples (blood and sputum ) collected will be considered a gift to the Oxford, and I understand that I will not derive personal or financial benefit beyond the explacompensation amount. | • | | |
| 6. | I agree to the genetic analysis of my samples, as detailed in the Participant Information Shee the results will not have implications for me personally. | t. I understand | | |
| 7. | I understand that my data may be shared with other researchers in a form that does not ider researchers may be outside of the UK. | ntify me. These | | |
| 8. | I agree to take part in this study. | | | |
| OPTIONAL - <u>The following are optional, answering "No" to any or all will not affect your ability to participate in the study.</u> | | | Yes | No |
| 9. | To avoid repeated testing, I agree that if I am not enrolled into this study and apply to enter another study conducted by the Jenner Clinical Vaccine Trials Group, my screening results may be used in that study, where appropriate. | | | |
| 10. | I agree that my contact details may be stored so that I may be informed of opportunities to p future vaccine related research. I understand that agreeing to be contacted does not oblige r participate in any further studies. | | | |
| Signe | d: Date: | | _ | |
| Name | e:(in block letters) Volunteer numbe | r <u>:</u> | _ | |

When completed, photocopy and provide 1 copy to the volunteer. Retain original for the research file.

\_\_\_\_\_ (in block letters)

Date: \_\_\_\_\_

Signature of Investigator:

Name of Investigator: \_\_\_